CLINICAL TRIAL: NCT05290688
Title: Cellular microRNA Signatures in Multiple Sclerosis
Acronym: SEP-MIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Pasteur (Industry)
Collaborators: Höpital La Pitié-Salpêtrière (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-044; 2021-A02983-3 (Other: ID-RCB)
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Inflammation; IFN-beta; Autoimmunity; Gene regulation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Inflammation; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: 20 untreated RRMS patients divided into 2 groups: 10 RRMS in relapsing phase 10 RRMS in relapse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Untreated RRMS patients (Other): Untreated RRMS patients with a 50 ml blood sample during their routine care
  Interventions: Genetic: 50 ml blodd sampling

INTERVENTIONS:
Genetic: 50 ml blodd sampling — 50 ml blood sampling for genetic analysis (expression profiles of microRNAs)

SUMMARY:
A limited number of studies on microRNA expression variation in immune cells have been reported in relapsing-remitting multiple sclerosis (RRMS). These studies have been performed mostly on a small scale and on whole blood mononuclear cells (PBMC).

In a number of cases, RRMS progresses to a severe secondary neurodegenerative form. In this context, it is important to look for biomarkers that could indicate the pathogenic activity of certain immune cell subpopulations.

DETAILED DESCRIPTION:
SEP-MIR is a prospective, single-center, descriptive study.

Participants will be recruited among adult patients with RRMS coming for a follow-up consultation in the Neurology Department, Nervous System Diseases Pole, at the hôpital Pitié - Salpêtrière (Paris).

As this is a descriptive study, the recruitment of 20 participants (10 patients with relapsing-remitting MS and 10 patients with relapsing-remitting MS) should meet the objectives of this study.

A 50 ml blood sample will be obtained from each participant and several clinical data regarding their pathology will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian population
* Female and male individuals with an f/m ratio of 2-4/1
* Individuals with RRMS according to the 2010 McDonald criteria for less than 15 years, with EDSS 1-6, in remission or relapse
* Participant's condition compatible with a maximum of 50 ml of blood collection
* Persons affiliated with a social security plan.

Exclusion Criteria:

* MS treatment with steroidal anti-inflammatory drugs, immunomodulators or immunosuppressants within 2 months prior to blood collection
* Persons with acute and chronic infectious disease, autoimmune/inflammatory disease or cancer other than MS
* Pregnant or lactating women
* Be under guardianship,
* Be deprived of liberty by judicial or administrative decision, or be under legal protection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
microRNA expression profiles in immune cell populations from RRMS patients | 2 years
  RNAseq and/or Nanostring sequencing of PBMCs from RRMS patients

SECONDARY OUTCOMES:
microRNA expression profiles in unstimulated and stimulated CD4+ T cell populations ex vivo from RRMS patients | 2 years
  RNAseq and/or Nanostring sequencing of unstimulated and stimulated CD4+ T cell populations ex vivo from RRMS patients
microRNA expression profiles in monocytes from RRMS patients | 2 years
  RNAseq and/or Nanostring sequencing of monocytes from RRMS patients

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Michel, PhD, Study Director — Institut Pasteur
Locations (1):
- Hôpital La Pitié - Salpêtrière, Paris, France